CLINICAL TRIAL: NCT03990857
Title: Comprehensive Care Protocol in New Diagnosis of Type 2 Diabetes Mellitus and Associated Comorbidities in Primary Care: Quasi-experimental Study.
Brief Title: Comprehensive Care Protocol in New Diagnosis of Type 2 Diabetes Mellitus and Associated Comorbidities in Primary Care
Acronym: PICDM2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4R16/045
Record Dates: First submitted 2019-06-13; First posted 2019-06-19 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes
Keywords: comorbidities comprehensive care
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Primary Health Care

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Group of participants with a recent DM2 debut (less than 5 months) treated according to the comprehensive care protocol in DM2 with comorbidities attended in Primary care nurse office
  Interventions: Other: Comprehensive care protocol in new diagnosis of Type 2 Diabetes Mellitus and associated comorbidities in Primary Care
- comparison group (No Intervention): Participants in the study that do not receive the intervention. usual care.

INTERVENTIONS:
Other: Comprehensive care protocol in new diagnosis of Type 2 Diabetes Mellitus and associated comorbidities in Primary Care — This comprehensive intervention is developed in a structured way in the Primary care nurse office. 5 individual intensive visits will be carried out with a weekly or bi-weekly frequency (according to the learning process) to work for an integral care and to transmit the knowledge and skills required. The maximum time expected to receive this 5 visits is 3 months. At least one of the visits, preferably the one that deals with dietary aspects, the patient is asked to be visited with the partner, child or cohabiting person. The research team elaborated the support material with the minimum contents that every patient that begins with T2DM and other chronic pathologies should know. It allows incorporating cultural and emotional aspects. It was agreed with hospital diabetes educators and family doctors. A graphic designer gave an enticing design. A group of patients verified their utility and intelligibility. It is delivered to the person and discussed during the intensification.
  Arms: Intervention

SUMMARY:
Introduction

Type 2 Diabetes is a very prevalent chronic disease in our environment. It usually exists with other chronic diseases. Although drug intensification at the time of new diagnosis has proven effective in reduction of cardiovascular and diabetes control and complications, an intensification of comprehensive health education has not been proven so. Currently, there is a great variability in practices of Primary Care nurses in front of the health education in the moment of new diagnosis.

The aim of this study is to evaluate the effectiveness of a systematic protocol with an integrated care in people with newly diagnosed type 2 diabetes (DM2) and associated comorbidities, which included 5 structured individual visits post-diagnosis with the Primary care nurse.

Methods

Quasi-experimental design, comparing a group of individuals taking part in the intervention with a similar group receiving usual care. Data will be collected at the beginning, at the end of the intervention and after 6 and 12 months. 10 primary care centers in the city of Barcelona will be selected on a convenience basis as IG and CG. The subjects of the GC will be monitored as usual. Performed analysis will be the baseline comparability between GI and GC in relationship to different variables as well as the changes in dependent variables along the study; establishing comparisons between GC and GI . The results will be measured in terms of quality of life related to health, development of biological parameters (HbA1c and weight) and compliance with the therapeutic plan.

Discussion

The results of this study will help to 1)demonstrate that by intensifying the hygienic-dietetic measures in the initial stage of DM2 diagnosis, the disease and associated co-morbidities are controlled in a better way. 2) validate a material that allows to decrease the variability in the care offered by primary care nurses to people in this group.

DETAILED DESCRIPTION:
Objectives

To evaluate the effectiveness of the systematic application of the comprehensive care protocol in people who debut in DM2 and associated comorbidities, applied during 3 months in primary care, in terms of quality of life related to Health, weigh loss and Glycosylated hemoglobin (HbA1c) compared to people who receive normal practice.

Secondary: To evaluate the effectiveness of the systematic application of the comprehensive care protocol of DM and associated comorbidities, during 3 months in primary care, in the parameters:

* Evolution of the specific biological parameters: TA, BMI, lipid profile, abdominal perimeter.
* Evolution of the consumption of drugs.
* Compliance with dietary recommendations.
* Increase in physical activity.
* Satisfaction / opinion of the participants. According to a questionnaire of user satisfaction of the ICS adapted to our study.
* Health frequentation in Primary Care Centers.

Methods and Analysis Study Design: A quantitative quasi-experimental design, multicenter, one-year follow-up, comparing a group of patients with a recent DM2 debut (less than 5 months) treated according to the comprehensive care protocol in DM2 with comorbidities, the intervention (IG), with a group of similar characteristics who receive the usual care (CG). The response variables will be evaluated before starting the care according to protocol, after (3 months) and at 6 and 12 months of initiating the intervention, in both groups.

Scope of the study: It will be developed in 10 urban primary care health centers, in 5 centers the intervention will be carried out and in 5 the controls will be selected. The allocation of a center as an intervention or comparison will be random. In the calculation of the sample the cluster effect attributable to this design has been considered.

Subjects of the study: The study population will consist of patients attended in the selected Primary Care Centers with a new diagnosis of DM2 (less than 5 months from the debut) that present comorbidity with an other chronic cardiovascular condition (Hypertension, dyslipidemia and/or obesity). Will be excluded COPD and IC, because they are attended with a specific protocol of care.

ELIGIBILITY:
Inclusion Criteria:

* People between both sexes between 18 and 80 years old with a recent (less than 5 months)diagnosis of DM 2 + comorbidity , assigned to the nurses that participate in the study and who give their consent to participate.

Exclusion Criteria:

* People who participate in a similar project.
* People with difficulty maintaining their participation for 12 months.
* People who have difficulty understanding and expressing themselves in Catalan or Spanish.
* People who have serious health problems: serious mental disease, terminal processes.
* People with COPD and IC, because they were included in another study with a specific care plan.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change is being assessed in Health Related Quality of Life will be measured through the EuroQoL (EQ-5D) | The outcome measure will be measured before, up to 3,6 and 12 months to assess its change
  The EQ-5D health questionnaire provides a simple descriptive profile and a single index value for health status.
HbA1c | up to 12 months.
  Glycosylated hemoglobin for having a clinical response.
Change is being assessed in Weigh | The outcome measure will be measured before, up to 3,6 and 12 months to assess its change
  Weigh for having a clinical response.

SECONDARY OUTCOMES:
Dietary habits: PREDIMED | baseline, up to 3,6 and 12 months.
  with the Predimed questionnaire. It consists of 14 questions. If the answer corresponds to a healthy practice, 1 point per question is counted. The range of answers goes from 0 (worst result) to 14 (best result).
Physical activity: IPAQ | baseline, up to 3,6 and 12 months.
  with the IPAQ questionnaire. The IPAQ asks about the exercise performed the last 7 days. It is structured to provide walking scores, moderate and high intensity activities. The final score of the short form requires the sum of the duration (in minutes) and frequency (days). The data obtained by the IPAQ can be shown as a continuous variable, for this each activity is measured by its energy requirements defined as MET's and in that way can be expressed in MET's-minute. More METs correspond to more exercise. Higher values represent a better outcome.
Use of services in the last year | Measure the year after diagnosis in both groups
  (Primary Care visits). Number or visits in GP and nurse office and at home during the year of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut català de la salut, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The derived data supporting the findings of this study will be available from the corresponding author [CL] on request.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Lapena C, Borras E, Digon C, Aznar R, Del Val Garcia JL, Castelblanco E, Garaikoetxea A, Laguna V. Effectiveness of a comprehensive care protocol in patients with new diagnoses of type 2 diabetes mellitus and associated comorbidities in primary care: study protocol of a quasi-experimental trial. BMJ Open. 2020 Jun 23;10(6):e033725. doi: 10.1136/bmjopen-2019-033725. PMID 32580980